CLINICAL TRIAL: NCT05978271
Title: An Observational Study Investigating the Experience of Patients Undergoing Active Insomnia Clinical Trials
Brief Title: Appraising Clinical Trial Experiences of Patients With Insomnia
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 81875001
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Insomnia
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Medical research participation percentages haven't always been fully representative of a given demographic.

The goal is to find out which aspects of a clinical trial may make it more difficult for patients to take part or see it through.

The data will be evaluated through different demographic lenses and identify trends that could help improve the experience of future insomnia patients during clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed.
* Participant has a diagnosis of insomnia.
* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.

Exclusion Criteria:

* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent.
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug(s) administration or interfere with the interpretation of safety results.
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with insomnia who are actively considering involvement in an observational clinical research, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in an insomnia clinical research. | 3 months
Number of insomnia patients who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: MichaelB B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yin X, Li W, Liang T, Lu B, Yue H, Li S, Zhong VW, Zhang W, Li X, Zhou S, Mi Y, Wu H, Xu S. Effect of Electroacupuncture on Insomnia in Patients With Depression: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2220563. doi: 10.1001/jamanetworkopen.2022.20563. PMID 35797047
- [Background] Liang X, Wang Q, Jiang Z, Li Z, Zhang M, Yang P, Wang X, Wang Y, Qin Y, Li T, Zhang T, Wang Y, Sun J, Li Y, Luo H, Li L. Clinical research linking Traditional Chinese Medicine constitution types with diseases: a literature review of 1639 observational studies. J Tradit Chin Med. 2020 Aug;40(4):690-702. doi: 10.19852/j.cnki.jtcm.2020.04.019. PMID 32744037
- [Background] Anand S, Tong H, Besag FMC, Chan EW, Cortese S, Wong ICK. Safety, Tolerability and Efficacy of Drugs for Treating Behavioural Insomnia in Children with Attention-Deficit/Hyperactivity Disorder: A Systematic Review with Methodological Quality Assessment. Paediatr Drugs. 2017 Jun;19(3):235-250. doi: 10.1007/s40272-017-0224-6. PMID 28391425

DOCUMENTS (1):
  • Informed Consent Form (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT05978271/ICF_000.pdf